CLINICAL TRIAL: NCT06071845
Title: Assessment of a Minimally Invasive Collection Device for Molecular Analysis of Esophageal Samples for the Non-endoscopic Detection of Barrett's Esophagus With and Without Dysplasia
Brief Title: Assessment of a Minimally Invasive Collection Device for Molecular Analysis of Esophageal Samples
Acronym: SOS4C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-010506; NCI-2023-07131 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Barretts Esophagus With Dysplasia; Barrett's Esophagus Without Dysplasia; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: Prospective multi-center case control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Known or Suspected Barrett's Esophagus (Case Arm) (Experimental): Investigators will follow Cytosponge Cell Collection Kit Instructions for Use to administer and retrieve the Cytosponge device.c. After the sponge is retrieved, it will then be placed in a vial of cell preservative solution (PN DD-13631, Exact Sciences, Madison, WI) and shipped to the Exact Sciences laboratory for further processing and subsequent analysis.
  Interventions: Device: Cytosponge Procedure; Diagnostic Test: Endoscopic Assessment
- No Known Barrett's Esophagus (Control Arm) (Active Comparator): Participants will undergo a diagnostic clinically indicated sedated endoscopy with standard endoscopic equipment.
  Interventions: Device: Cytosponge Procedure; Diagnostic Test: Endoscopic Assessment

INTERVENTIONS:
Device: Cytosponge Procedure — Investigators will follow the Cytosponge Cell Collection Kit Instructions for Use to administer and retrieve the Cytosponge device.
Diagnostic Test: Endoscopic Assessment — Participants will undergo a diagnostic clinically indicated sedated endoscopy with standard endoscopic equipment.

SUMMARY:
This clinical trial evaluates the use of cytosponge, a minimally invasive collection device, for the detection of Barrett's esophagus (BE) in patients undergoing endoscopy. Non-endoscopic swallowable encapsulate sponge cell collection devices combined with markers for BE/esophageal adenocarcinoma (EAC) detection are a guideline-endorsed alternative to endoscopy for BE screening. The Oncoguard registered trademark Esophagus test (OGE) test uses esophageal cytology specimens collected with a minimally invasive, non-endoscopic, encapsulated sponge sampling device to identify BE/EAC biomarkers that indicate whether a patient should undergo diagnostic endoscopy. The OGE test is a simple and cost effective screening method that may lower barriers to widespread adoption of BE screening in at risk patients, resulting in increased and earlier detection of BE/EAC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure Deoxyribonucleic acid (DNA) yield from esophageal cytology samples collected with the Cytosponge device.

II. Evaluate the methylated DNA markers (MDM) levels and accuracy of the Oncoguard Esophagus test (OGE test) for the detection of methylated DNA markers in Cytosponge collected esophageal cytology samples.

SECONDARY OBJECTIVES:

I. Assess the tolerability of the Cytosponge device using a tolerability questionnaire II. Evaluate presence of any trauma to the esophagus from the passage of the Cytosponge device using the endoscopic injury score.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients with known or suspected Barrett's Esophagus undergo a biopsy and sample collection with the cytosponge followed by standard of care endoscopy and complete surveys while on study.

ARM II: Patients without known or suspected Barrett's Esophagus undergo a biopsy and sample collection with the cytosponge followed by standard of care endoscopy and complete surveys while on study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known or suspected Barrett's esophagus (BE) (cases)

  * Patients between the ages of 18-90.
  * Patients with a BE segment ≥ 1cm in maximal extent endoscopically or suspected BE in medical record.
  * Histology showing evidence of intestinal metaplasia with or without presence of dysplasia or suspected BE in medical record.
  * Undergoing clinically indicated endoscopy.
* Subjects without known history of BE (controls)

  * Undergoing clinically indicated diagnostic endoscopy

Exclusion Criteria:

* For subjects with or without known evidence of BE (on history or review of medical records)

  * Pregnant or lactating females.
  * Patients who are unable to consent.
  * Patients with current history of uninvestigated dysphagia.
  * History of eosinophilic esophagitis, achalasia.
  * Patients on oral anticoagulation including Coumadin, Warfarin.
  * Patients on antiplatelet agents including Clopidogrel, unless discontinued for three to five days prior to the Cytosponge procedure.
  * Patients on oral thrombin inhibitors including Dabigatran and oral factor Xa inhibitors such as rivaroxaban, apixaban and edoxaban, unless discontinued for three to five days prior to the Cytosponge procedure.
  * Patients with history of known esophageal or gastric varices or cirrhosis.
  * Patients with history of surgical esophageal resection for esophageal carcinoma.
  * Patients with congenital or acquired bleeding diatheses.
  * Patients with a history of esophageal squamous dysplasia.
  * Patient has known carcinoma of the foregut (pancreatic, bile duct, ampullary, stomach, or duodenum) within 5 years prior to study enrollment.
  * Patient has received chemotherapy class drugs or radiation to treat mediastinal or esophageal cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
DNA yield from esophageal cytology samples collected with the Cytosponge device | 12 months
  DNA concentration from samples collected with the Cytosponge device will be compared with DNA concentration previously observed from samples collected with the EsophaCap device on another study. The DNA concentration range for EsophaCap collected specimens ranged from 0.4 to 285ng/uL.
Accuracy of the Oncoguard Esophagus (OGE) test | 12 months
  Methylated DNA marker (MDM) levels and accuracy (sensitivity and specificity) will be evaluated to determine the accuracy of the OGE test using Cytosponge-collected esophageal samples. Accuracy will be established using upper endoscopy with pathology confirmed histology as the criterion standard for the diagnosis of Barrett's Esophagus (BE). The recently established algorithm for defining the OGE test as positive or negative (from EsophaCap samples collected from another study) will be utilized to adjudicate the Cytosponge samples as positive or negative. Accuracy of the OGE test for the Cytosponge device will be assessed in relation to the estimates and confidence intervals previously observed.

SECONDARY OUTCOMES:
Tolerability of the Cytosponge device | 7 days
  Tolerability will be assessed with a 6-question Tolerability Questionnaire using a 0-10 pain scale where 0 is none and 10 is severe (0 is good and 10 is not good).
Trauma to the esophagus from the passage of the Cytosponge device | 7 days
  Presence of any trauma from the passage of the sponge will be assessed and recorded photographically during the sedated endoscopy. This will be defined as: No evidence of trauma; Superficial mucosal abrasion without bleeding; Superficial mucosal tear abrasion with minimal oozing similar to that from biopsy; Deep mucosal abrasion without bleeding; Deep mucosal abrasion with greater than minimal oozing; or Bleeding requiring endoscopic therapy or perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Prasad G. Iyer, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (5):
- United States (5):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Long Island Jewish Medical Center | Northwell Health, New Hyde Park, New York

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials